CLINICAL TRIAL: NCT01823900
Title: A Randomized, Open Label, Single-Dose, 2-Way Cross-over Clinical Trial to Compare the Safety and Pharmacokinetic Characteristics of Combination of Rosuvastatin and CS-866 and DWJ1276 in Healthy Male Volunteers
Brief Title: Safety and Pharmacokinetic Comparison of Co-administration and a Combination Drug of Rosuvastatin and Olmesartan in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, Kyungsoo Park, Associate Professor, Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DWJ1276
Record Dates: First submitted 2013-03-24; First posted 2013-04-04 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
Keywords: Pharmacokinetics

ARMS (1):
- Test and reference formulations (Experimental): Test formulation and reference formulation given orally 7 days apart in a fasted state
  Interventions: Drug: Test formulation; Drug: Reference formulation

INTERVENTIONS:
Drug: Test formulation — Single administration of a combination tablet of Rosuvastatin 20mg and Olmesartan 40mg
Drug: Reference formulation — Co-administration of Rosuvastatin 20mg tablet and Olmesartan 40mg tablet

SUMMARY:
This study investigates safety and pharmacokinetic comparison of DWJ1276, a combination drug of Rosuvastatin and Olmesartan (test formulation), and co-administration of Rosuvastatin and Olmesartan (reference formulation) for single dose in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers between the ages of 20 and 50 and within 20% of their ideal body weight, without congenital abnormality or chronic disease

Exclusion Criteria:

* History of cardiovascular, pulmonary, renal, endogenous, gastrointestinal, hematologic, neurologic or hemorrhagic disease;
* Clinically significant findings on routine laboratory (hematology, serum chemistry and urinalysis) or ECG tests;
* Use of prescription drugs in the 14 days immediately prior to starting the study that had the potential to interact with the study medication;
* Use of any substance that could induce or inhibit drug metabolism enzymes

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2012-01; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Profile of Pharmacokinetics | 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72 hours post-dose
  Cmax, Area Under Curve (0 to last sampling time)

SECONDARY OUTCOMES:
Profile of Pharmacokinetics | 0, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72 hours post-dose
  Tmax, Area Under Curve (0 to infinity), T_1/2

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Son H, Roh H, Lee D, Chang H, Kim J, Yun C, Park K. Pharmacokinetics of rosuvastatin/olmesartan fixed-dose combination: a single-dose, randomized, open-label, 2-period crossover study in healthy Korean subjects. Clin Ther. 2013 Jul;35(7):915-22. doi: 10.1016/j.clinthera.2013.05.016. Epub 2013 Jun 27. PMID 23810276